CLINICAL TRIAL: NCT06869265
Title: A Multicenter, Single-Arm, Prospective Clinical Study of Thiotepa Combined With Busulfan and Fludarabine Conditioning Regimen for Haploidentical Hematopoietic Stem Cell Transplantation in Elderly Patients With High-Risk Acute Myeloid Leukemia
Brief Title: Thiotepa Combined With Busulfan and Fludarabine Conditioning Regimen for Haploidentical Hematopoietic Stem Cell Transplantation in Elderly Patients With High-Risk Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHD035-001
Record Dates: First submitted 2025-03-02; First posted 2025-03-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia (AML); High Risk Acute Myeloid Leukemia(AML); Relapsed/Refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- thiotepa 5 mg/kg/day ; busulfan 3.2 mg/kg/day ; fludarabine 30 mg/m²/day (Experimental): Eligible patients will receive the following conditioning regimen: thiotepa 5 mg/kg/day on Days -10 to -9; busulfan 3.2 mg/kg/day on Days -8 to -6; fludarabine 30 mg/m²/day on Days -6 to -2; and rabbit anti-thymocyte globulin (rATG) 1.5-2.5 mg/kg/day on Days -5 to -2. Hematopoietic stem cell infusion will be performed on Day 0. Graft-versus-host disease (GVHD) prophylaxis will include cyclosporine A (CsA), mycophenolate mofetil (MMF), and methotrexate (MTX).
  Interventions: Drug: Thiotepa ;busulfan;fludarabine

INTERVENTIONS:
Drug: Thiotepa ;busulfan;fludarabine — Eligible patients will receive the following conditioning regimen: thiotepa 5 mg/kg/day on Days -10 to -9; busulfan 3.2 mg/kg/day on Days -8 to -6; fludarabine 30 mg/m²/day on Days -6 to -2; and rabbit anti-thymocyte globulin (rATG) 1.5-2.5 mg/kg/day on Days -5 to -2. Hematopoietic stem cell infusion will be performed on Day 0. Graft-versus-host disease (GVHD) prophylaxis will include cyclosporine A (CsA), mycophenolate mofetil (MMF), and methotrexate (MTX).

SUMMARY:
Abstract:

This clinical study is designed to evaluate the efficacy and safety of a thiotepa, busulfan, and fludarabine (TBF) conditioning regimen for haploidentical hematopoietic stem cell transplantation (haplo-HSCT) in elderly patients (≥55 years) with high-risk acute myeloid leukemia (AML). A total of 56 eligible patients will be enrolled in this prospective, single-arm, multicenter trial.

Study Design:

This is a multicenter, single-arm, prospective clinical trial. Eligible patients will receive the following conditioning regimen: thiotepa 5 mg/kg/day on Days -10 to -9; busulfan 3.2 mg/kg/day on Days -8 to -6; fludarabine 30 mg/m²/day on Days -6 to -2; and rabbit anti-thymocyte globulin (rATG) 1.5-2.5 mg/kg/day on Days -5 to -2. Hematopoietic stem cell infusion will be performed on Day 0. Graft-versus-host disease (GVHD) prophylaxis will include cyclosporine A (CsA), mycophenolate mofetil (MMF), and methotrexate (MTX). The primary endpoint of this study is 1-year relapse-free survival (RFS).

Inclusion Criteria:

Age 55-70 years (inclusive). Diagnosis of high-risk AML , include relapsed/refractory AML or CR MRD+ or ELN22 adverse risk group .Relapsed/refractory AML defined as at least one of the following: recurrence of leukemia cells in peripheral blood or bone marrow blasts >5% after complete remission (CR), failure to achieve remission after two courses of standard induction therapy, relapse within 12 months after consolidation therapy, relapse after 12 months that is refractory to conventional chemotherapy, multiple relapses, or persistent extramedullary leukemia）.

Scheduled to undergo haploidentical hematopoietic stem cell transplantation (haplo-HSCT).

Adequate organ function. Eastern Cooperative Oncology Group (ECOG) performance status ≤2. Written informed consent obtained.

Exclusion Criteria:

Unwillingness or refusal to accept the study treatment protocol. Presence of donor-specific anti-HLA antibodies. Known human immunodeficiency virus (HIV) infection. Active hepatitis B or C, or chronic active hepatitis. Uncontrolled active infection at the time of enrollment. Any other condition deemed by the investigator as unsuitable for study inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-70 years (inclusive).
2. Diagnosis of high-risk AML , include relapsed/refractory AML or CR MRD+ or ELN22 adverse risk group . Relapsed/refractory AML defined as at least one of the following: recurrence of leukemia cells in peripheral blood or bone marrow blasts >5% after complete remission (CR), failure to achieve remission after two courses of standard induction therapy, relapse within 12 months after consolidation therapy, relapse after 12 months that is refractory to conventional chemotherapy, multiple relapses, or persistent extramedullary leukemia .
3. Scheduled to undergo haploidentical hematopoietic stem cell transplantation (haplo-HSCT).
4. Adequate organ function.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
6. Written informed consent obtained.

Exclusion Criteria:

1. Unwillingness or refusal to accept the study treatment protocol.
2. Presence of donor-specific anti-HLA antibodies.
3. Known human immunodeficiency virus (HIV) infection.
4. Active hepatitis B or C, or chronic active hepatitis.
5. Uncontrolled active infection at the time of enrollment.
6. Any other condition deemed by the investigator as unsuitable for study inclusion.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
1-year Relapse-Free Survival,（RFS） | 1-year

SECONDARY OUTCOMES:
1-year Overall Survival | 1-year
1-year Relapse Rate | 1-year
1-year Non-Relapse Mortality | 1-year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China